CLINICAL TRIAL: NCT03274895
Title: Randomized, Active-Controlled, Phase 3 Study to Evaluate Efficacy, Safety and Tolerability of 0.08% PHMB Ophthalmic Solution in Comparison With 0.02% PHMB + 0.1% Propamidine Combination Therapy in Subjects Affected by Acanthamoeba Keratitis
Brief Title: Polihexanide (PHMB) Eye Drops in Patients Affected by Acanthamoeba Keratitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SIFI SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 043/SI
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Results first posted 2023-08-02 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Acanthamoeba Keratitis
Keywords: polihexanide; propamidine; confocal microscopy
MeSH Terms: conditions — Acanthamoeba Keratitis | interventions — polihexanide; dibrompropamidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PHMB 0.08% plus placebo (Experimental): polihexanide (PHMB) 0.08% and placebo were administered in the affected eye until clinical resolution for a maximum of 12 months
  Interventions: Drug: PHMB 0.08%; Drug: placebo
- PHMB 0.02% plus propamidine 0.1% (Active Comparator): polihexanide (PHMB) 0.02% and propamidine 0.1% were administered in the affected eye until clinical resolution for a maximum of 12 months
  Interventions: Drug: Propamidine 0.1%; Drug: PHMB 0.02%

INTERVENTIONS:
Drug: PHMB 0.08% — 16 drops in a day in the affected eye for 5 days followed by 8 drops in a day for 7 days,6 drops in a day for 7 days and 4 drops in a day up to clinical resolution
  Other Names: Polihexanide 0.8 mg/ml
  Arms: PHMB 0.08% plus placebo
Drug: Propamidine 0.1% — 16 drops in a day in the affected eye for 5 days followed by 8 drops in a day for 7 days,6 drops in a day for 7 days and 4 drops in a day up to clinical resolution
  Other Names: Brolene eye drops
  Arms: PHMB 0.02% plus propamidine 0.1%
Drug: placebo — 16 drops in a day in the affected eye for 5 days followed by 8 drops in a day for 7 days,6 drops in a day for 7 days and 4 drops in a day up to clinical resolution
  Other Names: Brolene vehicle
  Arms: PHMB 0.08% plus placebo
Drug: PHMB 0.02% — 16 drops in a day in the affected eye for 5 days followed by 8 drops in a day for 7 days,6 drops in a day for 7 days and 4 drops in a day up to clinical resolution
  Other Names: Polihexanide 0.2 mg/ml
  Arms: PHMB 0.02% plus propamidine 0.1%

SUMMARY:
Prospective randomized study to evaluate the efficacy, safety and tolerability of 0.08% polihexanide (PHMB) eye drops in patients affected by acanthamoeba keratitis.

130 subjects were assigned to one of the following 2 treatment groups: Group 1: 0.08% polihexanide (PHMB) + placebo Group 2: 0.02% polihexanide (PHMB) + 0.1% propamidine

DETAILED DESCRIPTION:
This was a randomized, assessor-masked, active-controlled, multiple center, parallel-group phase 3 study to evaluate the efficacy, safety and tolerability of 0.08% polihexanide (PHMB) ophthalmic solution compared to the conventional 0.02% polihexanide (PHMB) + 0.1% propamidine in patients affected by acanthamoeba keratitis.

The study was designed as a superiority study with the possibility to test for non-inferiority if the superiority hypothesis was not met (CPMP/EWP/482/99).The study consisted of an eligibility screening visit, a treatment period including monthly follow-up visits until a clinical resolution was obtained (within a maximum of 1 year), followed by 2 post-treatment off-therapy visits (30 and 90 days after treatment discontinuation). 130 subjects with confirmed diagnosis of acanthamoeba keratitis (clinical signs plus positive confocal microscopy findings) were assigned to one of the following treatment groups in a ratio of 1:1.

Group 1: 0.08% PHMB + placebo Group 2: 0.02% PHMB + 0.1% propamidine

ELIGIBILITY:
Inclusion Criteria:

1. willing to give informed consent
2. man or woman of any race and ≥12 years of age
3. able to understand and willing to comply with study procedures, restrictions and requirements
4. Clinical findings consistent with Acanthamoeba keratitis
5. Confocal microscopy findings consistent with Acanthamoeba keratitis
6. The following previous treatments for Acanthamoeba keratitis are eligible: antibiotics, antiviral and antifungal drugs, antiinflammatory drugs
7. Females of childbearing potential will be included if they are either sexually inactive or using one highly effective contraceptive
8. Females of childbearing potential agree to remain sexually inactive or to keep the same birth control method for at least 28 days following the last study drug dose
9. A female of non-childbearing potential must have undergone one sterilization procedures at least 6 months prior to the first study drug dose
10. A non-vasectomized male subject agrees to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study drug and the female partner agrees to comply with inclusion 7 or 8. For a vasectomized male who has had his vasectomy 6 months or more prior to study start, it is required that they use a condom during sexual intercourse. A male who has been vasectomized less than 6 months prior to study start must follow the same restrictions as a non-vasectomized male.
11. If male, they must agree not to donate sperm from the first study drug dose until 90 days after dosing

Exclusion Criteria:

1. Subject with documented history and/or clinical signs of concomitant presence of an ocular infection caused by viruses (herpes simplex virus [HSV]) or fungi.
2. Subject treated with drugs having effects on Acanthamoeba cysts prior to study entry, including biguanides (PHMB, chlorhexidine) and diamidines (propamidine, hexamidine).
3. Subjects requiring systemic immunosuppression for Acanthamoeba associated scleritis.
4. Subjects requiring urgent surgical intervention for advanced Acanthamoeba keratitis in either eye (e.g., for advanced corneal thinning/melting etc.).
5. Subject with known or suspected allergy to biguanides, diamidines or intolerance to any other ingredient of the investigational treatments.
6. Subject affected by immunodeficiency diseases or taking systemic immunosuppressive therapy.
7. Subject with a major systemic disease or other illness that would, in the opinion of the investigator, compromise subject's safety or interfere with the collection or interpretation of study results.
8. If female, pregnancy, planned pregnancy, or breast-feeding
9. Subject is participating in another interventional clinical study with an experimental or unapproved/unlicensed therapy or has participated in another interventional clinical study within 4 weeks prior to this study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2017-08-13 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Dart, MD, Principal Investigator — Moorfield's Hospital London
Locations (6):
- Italy (2):
  - San Raffaele Hospital, Milan
  - San Giovanni and Paolo Hospital, Venice
- University Clinical Center Medical University of Silesia, Katowice, Poland
- United Kingdom (3):
  - Moorfields Hospital, London
  - Manchester Royal Eye Hospital, Manchester
  - University Hospital Southampton, Southampton

REFERENCES:
- [Background] Papa V, Rama P, Radford C, Minassian DC, Dart JKG. Acanthamoeba keratitis therapy: time to cure and visual outcome analysis for different antiamoebic therapies in 227 cases. Br J Ophthalmol. 2020 Apr;104(4):575-581. doi: 10.1136/bjophthalmol-2019-314485. Epub 2019 Aug 10. PMID 31401556
- [Background] Papa V, van der Meulen I, Rottey S, Sallet G, Overweel J, Asero N, Minassian DC, Dart JKG. Safety and tolerability of topical polyhexamethylene biguanide: a randomised clinical trial in healthy adult volunteers. Br J Ophthalmol. 2022 Feb;106(2):190-196. doi: 10.1136/bjophthalmol-2020-317848. Epub 2020 Nov 25. PMID 33239413
- [Derived] Dart JKG, Papa V, Rama P, Knutsson KA, Ahmad S, Hau S, Sanchez S, Franch A, Birattari F, Leon P, Fasolo A, Kominek EM, Jadczyk-Sorek K, Carley F, Hossain P, Minassian DC. The Orphan Drug for Acanthamoeba Keratitis (ODAK) Trial: PHMB 0.08% (Polihexanide) and Placebo versus PHMB 0.02% and Propamidine 0.1. Ophthalmology. 2024 Mar;131(3):277-287. doi: 10.1016/j.ophtha.2023.09.031. Epub 2023 Oct 5. PMID 37802392

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from August 2017 and March 2021. Of the 135 enrolled participants 134 were randomized to treatment
Groups:
- PHMB 0.08% Plus Placebo; PHMB 0.02% Plus Propamidine 0.1%: 16 drops of each solution in a day for 5 days,8 drops each in a day for 7 days,6 drops each in a day for 7 days and 4 drops each in a day up to clinical resolution
Period: Overall Study
Arm/Group | PHMB 0.08% Plus Placebo | PHMB 0.02% Plus Propamidine 0.1%
Started | 69 (3 patients had no confirmation of diagnosis and therefore the overall number of participants analyzed is 66) | 65 (4 patients had no confimation of diagnosis and therefore the overall number of participants analyzed is 61)
Completed | 56 | 54
Not Completed | 13 | 11
Not completed — Lack of Efficacy | 1 | 0
Not completed — Adverse Event | 8 | 7
Not completed — Lost to Follow-up | 1 | 0
Not completed — Diagnosis not confirmed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PHMB 0.08% Plus Placebo | PHMB 0.02% Plus Propamidine 0.1% | Total
Number analyzed (Participants) | 69 | 65 | 134
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [25 to 43] | 36 [26 to 49] | 35 [25 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 37 | 78
  Male | 28 | 28 | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Visual acuity (best corrected) [Median (Inter-Quartile Range); unit: LogMAR] | 0.350 [0.150 to 0.70] | 0.260 [0.100 to 0.480] | 0.300 [0.150 to 0.700]
Culture positivity for Acanthamoeba [Count of Participants; unit: Participants] | 19 | 17 | 36
PCR positivity for Acanthamoeba [Count of Participants; unit: Participants] | 33 | 25 | 58

OUTCOME MEASURES:

1. Primary Outcome: Clinical Resolution Rate
Description: Percentage of patients cured 30 days after discontinuing all study therapies, within 12 months of randomization
Time Frame: 12 months
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PHMB 0.08% Plus Placebo | PHMB 0.02% Plus Propamidine 0.1%
Number analyzed (Participants) | 66 | 61
percentage of participants | 84.8 [73.9 to 92.5] | 88.5 [77.8 to 95.3]
Statistical Analysis 1: Comparison: PHMB 0.08% Plus Placebo vs PHMB 0.02% Plus Propamidine 0.1%; Test type: Non-Inferiority — Non-inferiority margin= 0.20; difference in proportion of resolution r = -0.036, 95% CI 2-sided [-0.154 to 0.081]

2. Secondary Outcome: Time to Cure
Description: Time needed to reach a clinical resolution
Time Frame: maximum 12 months
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | PHMB 0.08% Plus Placebo | PHMB 0.02% Plus Propamidine 0.1%
Number analyzed (Participants) | 66 | 61
days | 140 [117 to 150] | 114 [91 to 127]
Statistical Analysis 1: Comparison: PHMB 0.08% Plus Placebo vs PHMB 0.02% Plus Propamidine 0.1%; Test type: Other; p = 0.042, Log Rank

3. Secondary Outcome: Visual Acuity
Description: Final visual acuity (best corrected)
Time Frame: maximum 12 months
Population: Intent-to-treat
Measure: Median (Inter-Quartile Range); unit: LogMAR
Arm/Group | PHMB 0.08% Plus Placebo | PHMB 0.02% Plus Propamidine 0.1%
Number analyzed (Participants) | 66 | 61
LogMAR | 0.000 [0.000 to 0.250] | 0.000 [-0.080 to 0.150]
Statistical Analysis 1: Comparison: PHMB 0.08% Plus Placebo vs PHMB 0.02% Plus Propamidine 0.1%; Test type: Other; p = 0.577, ANCOVA

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | PHMB 0.08% Plus Placebo | PHMB 0.02% Plus Propamidine 0.1%
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/65
Other Adverse Events (participants affected / at risk) | 31/69 | 29/65
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PHMB 0.08% Plus Placebo (N=69) | PHMB 0.02% Plus Propamidine 0.1% (N=65)
eye pain (Eye disorders) | 9 (11) | 7 (7)
ocular hyperemia (Eye disorders) | 8 (9) | 7 (9)
lacrimation increased (Eye disorders) | 6 (6) | 2 (2)
conjunctival hyperemia (Eye disorders) | 2 (2) | 3 (4)
eye irritation (Eye disorders) | 1 (1) | 4 (4)
photophobia (Eye disorders) | 2 (2) | 3 (3)
eye inflammation (Eye disorders) | 3 (3) | 1 (3)
corneal epithelium defect (Eye disorders) | 3 (3) | 0 (0)
corneal infiltrates (Eye disorders) | 3 (3) | 0 (0)
eye pruritus (Eye disorders) | 1 (1) | 2 (2)
eye discharge (Eye disorders) | 2 (2) | 0 (0)
eye swelling (Eye disorders) | 2 (2) | 0 (0)
keratitis (Eye disorders) | 2 (2) | 0 (0)
ocular discomfort (Eye disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT03274895/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT03274895/SAP_001.pdf